CLINICAL TRIAL: NCT04388046
Title: Three-dimensional Evaluation of Pharyngeal Airway Measurements Following Class 2 Correction With Skeletally Anchored Herbst Appliance
Brief Title: Effect of Skeletally Anchored Herbst Appliance in Treatment of Skeletal Class 2 Due to Mandibular Retrusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khaled ELHabbak (Other)
Responsible Party: Sponsor-Investigator, Khaled ELHabbak, principal investigator, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 107
Record Dates: First submitted 2020-05-08; First posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Malocclusion, Angle Class II
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- skeletal class 2 malocclusion (Experimental): 10 patients treated with type IV Herbst appliance. The appliance was connected directly to the mandible by a bilateral reconstruction bone plates to provide a skeletal anchorage and avoid any mandibular teeth involvement
  Interventions: Device: Herbst fixed functional appliance

INTERVENTIONS:
Device: Herbst fixed functional appliance — Herbst appliance could be considered as an artificial joint working between maxilla and mandible. The appliance consists of a bilateral telescope mechanism attached to upper and lower jaws keeping the mandible in an anterior jumped position.

SUMMARY:
Ten adolescent female patients with Class 2 mandibular deficiency with a mean age of 16.5 ±1.71 years treated with type IV Herbst appliance.

Skeletally anchored appliance was connected directly to the mandible by a bilateral reconstruction bone plates to provide a skeletal anchorage, while connected to the maxilla through dental splint connecting upper canine, first premolar, first and second molars through the use of orthodontic bands connected together palatally by a heavy 1mm stainless steel wire.

The treatment duration was 9 months, then the appliances were removed,The Cone Beam Computed Tomography (CBCT) scans were taken before and immediately after Herbst treatment to analyse airway volume, also 3D measurement of the effective mandibular length has been taken. Cephalometric film was extracted from CBCT scans and analysed for dentoskeletal and soft tissue changes.

DETAILED DESCRIPTION:
The Herbst appliance was anchored by two reconstruction plates located bilaterally in the mandible between the canine and first premolar, while attached to the maxilla through dental splints utilizing orthodontic bands.

For each patient, two reconstruction plates were sent to the laboratory for LASER welding of the Herbst bases to the first hole of each reconstruction plate. This assembly was projected transmucosal and exposed into the oral cavity for direct connection with the Herbst appliance.

3D model for the mandible of each patient was printed with 3D printer machine after extracted from the patient CBCT.

The reconstruction plates were bended using a 3-jaw contouring and bending plier to be adapted to the printed model on the predetermined location between mandibular canine and 1st premolar bilaterally.Sterilization of the reconstruction plates were then preformed.

For surgical placement of reconstruction plates, An envelope flap with one releasing incision (three-corner flap)was made starting with the horizontal incision 3-mm apical to the gingival crest from the mesial surface of lower second premolar to the distal surface of lower lateral incisor on one side, then a vertical incision was made at the mesial end of the horizontal incision, extending apically to the chin level to allow unstrained placement of the reconstruction plate. The same procedures were performed on the other side.

Reconstruction plates were checked for proper positioning before fixation, the reconstruction plate was held in place, a small hole, only through the cortex of bone, was made by a surgical round bur through the middle hole of the reconstruction plate. This was followed by complete drilling using a surgical screw drill , a 2.3mm screw was used to fix the reconstruction plate in its place using the corresponding screwdriver .

Consequently, drilling of the upper and lower holes and fixation of screws were performed in the same manner, the same steps were performed to fix the contralateral reconstruction plate in its place.

The flaps were repositioned and sutured with 3/0 silk suture. Proper size readymade bands were selected for the maxillary first premolars, first and second molars, while canine bands were custom made specifically for each patient,The bands were accurately fitted in their place and an alginate impression for upper jaw was taken, washed and disinfected, then the bands were reinserted into the alginate impression and the impression was poured in white orthodontic stone. Then the cast was sent to the laboratory for constructing the palatal connecting wire and laser-welding the bands to the palatal wires. At this time, the bases of the telescopic mechanism were welded to the buccal surface of maxillary 1st molar bands.

In most patients, the mandible was advanced to an incisal edge-to-edge position in one step advancement, however, in two patients, because of the large overjet, the edge to edge position seemed to be traumatic, therefore two steps advancement about 5 mm each was undertaken using suitable spacers.

After adjustment and try in of all assembly, the maxillary splint was then cemented using glass ionomer cement .

The coupling heads of telescopic rods and tubes were secured inside the appliance bases on reconstruction plate and maxillary 1st molar bands respectively with the C-clip using plier.

Patients were recalled one day following appliance insertion then every two weeks.

The appliances were removed after nine months, the remnants of the glass ionomer cement were eliminated using finishing bur and teeth were polished using fluoride pumice powder with a rubber polishing cup in a low-speed hand piece. The reconstruction plates were removed with a second surgery.

Completion of orthodontic treatment for each patient was performed with fixed appliance to reach firm and functioning stable occlusion.

The images were acquired using CBCT machine. A scout view was obtained, and adjustments were made to ensure that all patients were correctly aligned in the scanner according to adjustment light beam before acquisition.

After acquisition, data were exported and transferred in digital imaging and communication in medicine (DICOM) format and downloaded via a CD to a personal computer for Airway volume calculation and extraction of both panoramic and lateral cephalometric radiograph using a specific software.

Serial steps were followed by the same investigator to standardize the measurements in all scans. An identification number was assigned to each CBCT image prior to measurement in order to mask the patient's name and the time point during CBCT analysis. The CBCT images were re-matched to the patient's name after data collection were completed.

The CBCT scans were taken before and immediately after Herbst treatment to analyze the following….

* 3D volumetric air way analysis.
* 3D measurement of the effective mandibular length.
* Cephalometric analysis after extraction from the CBCT. To ensure accurate and repeatable measures of all patients, all CBCT scans had to be oriented by the software before taking the measures.

ELIGIBILITY:
Inclusion Criteria:

* Skeletal and dental Class II malocclusion due to mandibular retrusion (SNB≤ 76° )
* Overjet ≥ 5.0 mm
* Normal or low FMA angle (≤ 28)
* Complete permanent dentition, excluding the third molars
* Minimum or no crowding in the mandibular arch
* All the patient involved in the study will be in stages 5 and 6 based on the modified cervical vertebral maturation stages (CVMS).

Exclusion Criteria:

* History of any medical problems that may interfere with orthodontic treatment
* Previous orthodontic treatment.
* Clinical signs and symptoms of temporomandibular disorders.
* Mandibular asymmetries.
* Bad oral hygiene.

Ages: 14 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2017-12-25 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2019-09-25 (Actual)

PRIMARY OUTCOMES:
three dimensional evaluation of pharyngeal airway volume | 9 months
  The air way analysis option was chosen to start the measurement. The nasopharynx, velopharynx, glossopharyngeal and the total air way horizontal boundaries all had been set parallel to Frankfort horizontal The vertical anterior boundary of pharyngeal airway was represented by the line perpendicular to FH plane and tangent to PNS.
  A quick method for determining the airway sensitivity has been chosen using a threshold value of 70 unit which was find optimum for airway segmentation.
  Consequently, the software was automatically converted the segmented airway into 3D volume.
  The 3D air way volume for the nasopharynx, velopharynx and glossopharyngeal as well as the total pharyngeal airway were calculated and tabulated.

SECONDARY OUTCOMES:
dento-skeletal changes | 9 months
  A constructed lateral cephalometric image was constructed from the patient's CBCT for assessment of maxillary and mandibular bony changes as well as the upper and lower anterior teeth.

CONTACTS AND LOCATIONS:
Overall Officials: khaled El-Habbak, Principal Investigator — Alazhar universty
Locations (1):
- Faculty of Dental Medicine, Al- Azhar University, Cairo-boys., Cairo, Egypt